CLINICAL TRIAL: NCT06730763
Title: Effect of Transcranial Direct Current Stimulation on Risk of Falling in Cerebral Palsy Spastic Hemiplegic Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dr. Ahmed Fathy Mahmoud Awd, Physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC.012/005208
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy (CP)
Keywords: cerebral palsy; spastic hemiplegia; risk of falling
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia | interventions — Transcranial Direct Current Stimulation; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): will receive selected traditional physical therapy program for improve balance and decrease risk of falling only.
  Interventions: Device: Transcranial direct current stimulation; Other: Exercise
- Group 2 (Active Comparator): will receive transcranial direct current stimulation plus selected traditional physical therapy program.
  Interventions: Other: Exercise

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation (TDCS) is a non-invasive, painless brain stimulation treatment that uses direct electrical currents to stimulate specific parts of the brain.
  Other Names: transcranial; TcDc
  Arms: Group 1
Other: Exercise — selected traditional physical therapy program for improve balance and decrease risk of falling
  Other Names: traditional

SUMMARY:
The purpose of this study was to determine:

* If there is an effect of transcranial direct current stimulation in improvement the functional balance in CP spastic hemiplegic children.
* If there are any changes in risk of falling in CP spastic hemiplegic children or not.

DETAILED DESCRIPTION:
With the decline of mobility comes a drastic increase in falling. However, people of all ages with cerebral palsy can fall easily due to imbalance issues and non-voluntary movements. Individuals with cerebral palsy (CP) can experience a variety of sensorimotor impairments that impact balance, making excessive tripping and falling among the most common concerns for ambulatory individuals with CP. Approximately 53-97% of ambulatory individuals fall at least once per year, causing injury, embarrassment, frustration, activity avoidance, and isolation. Although a study of over 1000 children found fall frequency was highest in gross motor function classification system (GMFCS) level II, research has not explored if this holds across the decades of adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 8-12 years old.
* Classified on levels II and III of the Gross Motor Function Classification System (GMFCS) (Palisiano et al.,1997).
* the ability to walk without the assistance of another individual for at least 12 months prior to the onset of the study, regardless of whether a gait-assistance device was needed (GMFCS level III) or not (GMFCS level II).
* (Pediatric Balance Scale, Timed Up and Go Test 'TUGT') and acceptance of the TDCS procedure.
* Ability to understand and follow simple instructions.
* Parent or guardian consent obtained

Exclusion Criteria:

* Orthopedic deformities, a history of surgery or neurolytic block in the previous 12 months,
* Diagnosis of epilepsy or having experienced convulsive crises (whether treated with medication or not) in at least the two years prior to the onset of the study, metal implants in the skull, or the use of hearing aids.
* Previous participation in a tDCS study within the past 6 months.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The Fall Risk test | From enrollment to the end of treatment at 8 weeks
  The fall risk test allowed identification of potential fall candidates. Test results were compared to age dependent normative data. Scores higher than normative values suggested more fall risk index

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided